CLINICAL TRIAL: NCT01082601
Title: Pulmonary Vein Isolation for Rhythm Control in Patients With Atrial Fibrillation and Left Ventricular Dysfunction: A Pilot Study
Brief Title: Catheter Ablation for Atrial Fibrillation and Heart Failure
Status: Withdrawn | Type: Observational
Why Stopped: no enrollment
Sponsor: St. Luke's-Roosevelt Hospital Center (Other)
Responsible Party: Sponsor
Other Study IDs: 09-137
Record Dates: First submitted 2010-03-05; First posted 2010-03-08 (Estimated); Last update posted 2012-10-17 (Estimated); Status verified 2011-06

CONDITIONS: Congestive Heart Failure; Atrial Fibrillation; Arrhythmia
Keywords: Catheter Ablation; Atrial Fibrillation; Congestive heart failure
MeSH Terms: conditions — Heart Failure; Atrial Fibrillation; Arrhythmias, Cardiac | interventions — Catheter Ablation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Optimal Medical therapy: Subjects with Class I,IIor III congestive heart failure on optimal medical therapy. Planned catheter ablation for paroxysmal or persistent atrial fibrillation. Paroxysmal AF defined as recurrent AF(2 or more episodes in one month) that terminate within seven days. Persistent AF defined as sustained beyond seven days, or lasting less than seven days but requiring pharmacologic or electrical cardioversion.
  Interventions: Procedure: Pulmonary Vein Isolation (PVI)

INTERVENTIONS:
Procedure: Pulmonary Vein Isolation (PVI) — Subjects with clinical indication for PVI, either paroxysmal or persistent AF failing medical management with rate or rhythm control medications.
  Other Names: Catheter Ablation

SUMMARY:
To compare heart function, symptoms, exercise capacity and quality of life in patients with Congestive Heart Failure (CHF) and Atrial Fibrillation (AF)before and after catheter ablation.

Hypothesis: Restoration and maintenance of sinus rhythm by catheter ablation, without the use of antiarrhythmic drugs, in AF and CHF improves heart failure status.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years to 80 years
* Clinical diagnosis of CHF based on symptoms (Shortness of breath, fatigue, peripheral edema)
* Systolic left ventricular dysfunction with ejection fraction 40% or less
* NYHA Class I, II or III heart failure
* Paroxysmal AF(2 or more episodes in one month) that terminate within 7 days:or persistent AF (more than 7 days or less than 7 days but terminated with pharmacologic or electrical cardioversion).
* Willing and able to sign informed consent

Exclusion Criteria:

* Previous ablation
* Left atrial size greater than 60mm(parasternal view on transthoracic echocardiogram)
* AF episodes triggered by another uniform arrhythmia(e.g.atrial flutter or atrial tachycardia)
* Active alcohol or drug abuse, which may be causative of AF
* Severe valvular disease requiring surgical repair
* Myocardial infarction within 6 months of enrollment
* Abnormality that prevents catheter introduction
* Coronary surgical revascularization or other cardiac surgery within 6 months of enrollment
* Patients in whom heart transplant expected with 6 months
* AF deemed secondary to a transient or correctable cause (e.g.electrolyte imbalance ,trauma,recent surgery,,infection, toxic ingestion or endocrinopathy
* Pregnancy or women of child bearing potential & not on reliable method of birth control
* Contraindication to Warfarin therapy or other bleeding diathesis
* Participation in another clinical trial
* Inaccessable to follow-up
* Life expectancy of less than 24 months caused by reasons other than heart disease
* Renal failure requiring dialysis
* Decompensated CHF within 48 Hours of enrollment
* Second or third degree AV block or sinus pause greater than 3 seconds, resting heart rate less 30 bpm without a permanent pacemaker
* A history of drug induced Torsades de Pointes or congenital long QT syndrome
* Currently responding to antiarrhythmic drug therapy
* Uninterrupted AF for more than 12 months prior to randomization unless sinus rhythm maintained for 24 hours or longer.
* Unwilling or unable to sign informed consent

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients seen in either the out patient or in hospital environment at St.Luke's-Roosevelt Hospital or The Valley Hospital, Ridgewood New Jersey, with systolic left ventricular dysfunction and atrial fibrillation. Class I-III CHF based on symptoms(shortness of breath,fatigue, peripheral edema and documented ejection fraction of less than 40%.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2010-04; Primary Completion 2012-01 (Actual); Study Completion 2012-01 (Actual)

PRIMARY OUTCOMES:
Improvement in LVESV by 15% or more from baseline at 6 months | 6 months

SECONDARY OUTCOMES:
Remodeling as demonstrated by atrial & ventricular dimensions on echocardiogram | 6 months
NYHA Class | 6 months
Quality of Life | 6 months
Six minute hall walk test | 6 months
Hospitalization for HF | one year
  Composite hospitalization for HF,thromboembolic complications, major bleeding or all cause mortality
Absence of Atrial fibrillation | one year

CONTACTS AND LOCATIONS:
Overall Officials: Suneet Mittal, MD, Principal Investigator — St. Luke's-Roosevelt Hospital Center
Locations (2):
- United States (2):
  - The Valley Hospital, Ridgewood, New Jersey
  - St.Luke's-Roosevelt Hospital, New York, New York